CLINICAL TRIAL: NCT07120516
Title: Co-creating School Community Intervention Program on Physical Activity to Increase Health Equity in Children and Adolescents
Acronym: Connection
Status: Recruiting | Type: Observational
Sponsor: Sandra Andrusaityte (Other)
Responsible Party: Sponsor-Investigator, Sandra Andrusaityte, associate professor, Vytautas Magnus University
Organization: Vytautas Magnus University (Other)
Other Study IDs: 2025 no. BE-2-27
Record Dates: First submitted 2025-07-30; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Obese Adolescents; Mental Health
Keywords: Child Health Inequalities; Physical Activity; Health Behavior in Adolescents
MeSH Terms: conditions — Psychological Well-Being; Motor Activity

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational and interventional study is to understand whether environmental and behavioral interventions can improve physical activity and health outcomes in children aged 12-16 years attending VDU Atžalynas Progymnasium, Lithuania.

The main questions it aims to answer are:

1. Does higher physical activity and improved lifestyle reduce health disparities among children living in disadvantaged social and economic conditions?
2. What is the relationship between environmental pollution, physical activity, and children's health indicators? Researchers will compare data from the cross-sectional group (baseline measurements only) and the intervention group (7-day activity tracking and follow-up after 3 months) to see if targeted environmental interventions improve children's physical activity, sleep quality, and health outcomes.

Participants will:

* Fill in questionnaires about health behaviors, well-being, and living environment (children and parents).
* Undergo physical measurements (blood pressure, height, weight, body composition).
* Wear a smart wristband for 7 days to monitor activity, sleep, and heart rate (only for selected participants).
* Attend a follow-up visit after 3 months (intervention group only).

DETAILED DESCRIPTION:
Non-communicable diseases (NCDs), such as cardiovascular diseases, obesity, and metabolic disorders, are a leading cause of morbidity and mortality worldwide. Evidence shows that insufficient physical activity, poor dietary habits, and exposure to environmental pollutants (such as PM2.5, PM10, and NO₂) significantly increase the risk of these conditions in children and adolescents. The negative impact of these risk factors is disproportionately higher in children living in socially and economically disadvantaged environments, perpetuating health inequalities from early life stages.

Physical activity and diet are modifiable risk factors. Interventions implemented at the community level, especially in school settings where children spend a large part of their day, have the potential to create long-term behavioral changes and reduce health disparities. However, the interaction between environmental exposures, social determinants, and physical activity on health outcomes is still poorly understood. There is a lack of comprehensive, evidence-based interventions targeting environmental and behavioral factors simultaneously in children from disadvantaged backgrounds.

The Connection Project is an international, multi-center observational and interventional study designed to:

* Assess the relationship between environmental exposures, physical activity, and health indicators in children aged 12-16 years.
* Implement and evaluate community-based environmental and behavioral interventions to promote healthier lifestyles.
* Contribute to evidence-based recommendations for reducing health inequities in school-age populations.

This study is supported by the European Commission under the ERA4Health program and funded nationally by the Research Council of Lithuania, in collaboration with multiple European research institutions in Portugal, Belgium, Spain, Lithuania, Latvia, Denmark, the Netherlands, and Italy.

Study Objectives

Primary Objectives:

1. To evaluate associations between environmental exposures (PM2.5, PM10, NO₂) and children's physical health indicators (blood pressure, body composition, anthropometrics).
2. To assess whether community-based environmental interventions can increase physical activity levels, improve sleep quality, and reduce disparities in health outcomes in disadvantaged populations.

Secondary Objectives:

1. To describe baseline health behaviors, dietary habits, and sleep patterns in children aged 12-16 years attending selected schools.
2. To assess parental perceptions of health, environmental exposures, and the built environment surrounding schools and homes.
3. To test the feasibility and acceptability of using CE-certified smart wristbands as objective tools for monitoring children's physical activity, sleep, and heart rate patterns over repeated measurement periods.
4. To provide recommendations for sustainable community-level interventions that can be scaled to other schools in Europe.

Study Design and Methodology: This is a two-phase study combining a cross-sectional baseline assessment and an in-depth interventional follow-up.

Phase 1 - Cross-Sectional Study: Population: Approximately 200 children aged 12-16 years attending *VDU Atžalynas Progymnasium in Kaunas, Lithuania.

* **Sampling:** Random selection from eligible students whose parents/legal guardians provide informed consent and who agree to participate.

Data Collection:

Questionnaires:

* Children: health behaviors, well-being, perceived environmental safety, dietary habits, physical activity frequency, sleep quality.
* Parents: social and demographic information, residential address for geocoding environmental exposure data.

Objective Measurements:

* Blood pressure (standardized automated device).
* Height and weight (stadiometer and calibrated scale).
* Body composition (bioelectrical impedance analysis). Environmental Exposure Data: Geocoded addresses will be linked with national air quality monitoring databases (PM2.5, PM10, NO₂) to estimate individual exposure levels.

All collected data will be pseudonymized and entered into secure electronic data capture systems. Each participant will be assigned a unique study ID to protect confidentiality.

Phase 2 - Interventional Study:

1. Population: Approximately 20 children (10% of Phase 1 participants) who consent to additional monitoring.
2. Intervention: Use of CE-certified smart wristbands for continuous 7-day monitoring of physical activity (step count, energy expenditure), sleep duration and quality, and heart rate variability.

Behavioral feedback will be provided to children and parents to encourage healthy routines. Community-level initiatives may include adjustments to the school environment (e.g., safe walking paths, organized activity breaks, improved playground access) to promote physical activity.

Timeline: Baseline monitoring (Visit 1): Placement of wristband, instructions provided (10 min). Day 7 (Visit 2): Retrieval of wristband, verbal feedback on experience (10 min). 3-Month Follow-Up (Visit 3): Repeated health measurements and 7-day monitoring period to assess changes in activity, sleep, and health indicators.

The goal is to evaluate feasibility, adherence, and preliminary health impact of combining environmental and behavioral interventions.

Data Management and Analysis: Personal identifiers will be kept separate from research data. Electronic files will be encrypted and stored on password-protected servers at Vytautas Magnus University. Access will be limited to authorized study staff. Data will be retained for 5 years after project completion before secure destruction.

Statistical Analysis:

1. Descriptive statistics for baseline health and environmental exposures.
2. Multivariate regression models to assess associations between pollution exposure, physical activity, and health outcomes.
3. Longitudinal comparisons (baseline vs. 3-month follow-up) to evaluate intervention effects.
4. Sensitivity analyses to account for missing data and confounding factors (e.g., socioeconomic status, age, sex).

Ethical Considerations: The study has been reviewed and approved by the Kaunas Regional Biomedical Research Ethics Committee.

Participation is voluntary; informed consent from parents/legal guardians and assent from children will be obtained prior to enrollment.

Participants may withdraw at any time without consequences. All procedures are non-invasive and involve minimal risk, limited to mild discomfort from measurements or wearing a wristband.

No compensation is provided; participation is voluntary and free of charge. Data confidentiality will be protected according to GDPR and national laws.

Expected Outcomes and Impact: The Connection Project is expected to:

* Provide new evidence on links between environmental pollution, physical activity, and health indicators in children.
* Demonstrate the feasibility of using wearable technologies for pediatric population health monitoring in community settings.
* Inform local and European public health policies aimed at reducing environmental and social determinants of health inequalities.
* Support future large-scale interventions to promote equitable access to physical activity opportunities and healthier lifestyles in disadvantaged youth populations.

International Collaboration: This project is part of a European consortium with research partners in: Portugal: University of Porto, Institute of Public Health; Belgium: Ghent University; Spain: ISGlobal, Barcelona; Latvia: Riga Stradins University; Denmark: University of Copenhagen; Netherlands: Amsterdam Public Health Research Institute and Italy: University of Turin

ELIGIBILITY:
Inclusion Criteria:

* Children aged 12-16 years
* Attending VDU Atžalynas Progymnasium (Kaunas, Lithuania)
* Written informed consent from parents/legal guardians and assent from the child
* Willingness to participate in questionnaires, physical measurements, and (if selected) wearable device monitoring

Exclusion Criteria:

* Younger than 12 or older than 16 years
* No signed informed consent from parents/legal guardians or refusal by the child
* Medical or psychological conditions that may interfere with participation (e.g., severe cardiovascular disease, mobility impairments, skin allergies preventing wearable use)

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population will consist of children aged 12-16 years enrolled in VDU Atžalynas Progymnasium (Kaunas, Lithuania). Participants will be selected from a general school population, with priority given to inclusion of children living in socially and economically disadvantaged environments. Eligible participants will be healthy volunteers without medical conditions that could interfere with the study procedures. Both parental consent and child assent are required for participation.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Change in systolic and diastolic blood pressure in children aged 12-16 years | Baseline (Day 0) and 3 months after intervention
  This outcome assesses changes in systolic and diastolic blood pressure (measured in mmHg) in participating children. Blood pressure will be measured using calibrated, CE-certified devices to evaluate the effect of increased physical activity and improved environmental conditions on cardiovascular health.
Change in body composition indicators in children aged 12-16 years | Baseline (Day 0) and 3 months after intervention
  This outcome includes changes in body mass index (BMI), fat mass percentage, weight (kg), and height (m). Measurements will be collected using validated, CE-certified body composition analyzers to assess improvements in physical health related to the intervention.

SECONDARY OUTCOMES:
Change in physical activity levels in children aged 12-16 years | Baseline (Day 0) and 3 months after intervention
  Assesses change in average daily step count and active minutes using CE-certified smart wristbands worn for 7 consecutive days. The data will reflect children's habitual physical activity levels before and after the intervention.
Change in self-reported well-being in children aged 12-16 years | Baseline (Day 0) and 3 months after intervention
  Assesses well-being using the KIDSCREEN-10 Index (range: 10-50; higher scores indicate better well-being). Children complete the validated questionnaire at each time point to capture psychological and social well-being changes post-intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Vytautas Magnus university, faculty of Natural Sciences, Environmental sciences, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided
De-identified individual participant data (IPD) collected during this study (questionnaire responses, anthropometric measurements, body composition, physical activity, and sleep monitoring data) may be shared with qualified researchers upon reasonable request for purposes of scientific validation, secondary analyses, and meta-analyses, in compliance with GDPR and national data protection laws. Data will be coded to protect participant identity and shared only after Ethics Committee approval and a signed data use agreement.

DOCUMENTS (3):
  • Study Protocol (2024-11-20): https://cdn.clinicaltrials.gov/large-docs/16/NCT07120516/Prot_000.pdf
  • Informed Consent Form: Informed consent form (parents) (2025-01-22): https://cdn.clinicaltrials.gov/large-docs/16/NCT07120516/ICF_001.pdf
  • Informed Consent Form: Informed consent form (children) (2025-01-22): https://cdn.clinicaltrials.gov/large-docs/16/NCT07120516/ICF_002.pdf